CLINICAL TRIAL: NCT01221519
Title: Randomized, Open, 4-way Crossover, Single Center, Phase I Relative Bioavailability Study in Type 2 Diabetes Mellitus Patients to Measure the Extent and Rate of Absorption of AZD1656 From Different Tablet Formulations
Brief Title: A Relative Bioavailability Study Measuring the Extent and Rate of Absorption of Different Tablet Formulations of AZD1656 in Type 2 Diabetes Mellitus (T2DM) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1020C00033
Record Dates: First submitted 2010-10-12; First posted 2010-10-15 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes Mellitus; High Blood Sugar
Keywords: Phase I; Bioavailability; Type 2 Diabetes Mellitus; Diabetic treatment; Metformin; High blood sugar
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — AZD1656

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 2 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 3 (Experimental): AZD1656
  Interventions: Drug: AZD1656

INTERVENTIONS:
Drug: AZD1656 — 3 different formulations, A, B and C of AZD1656 assessed before food intake and formulation B also after food intake

SUMMARY:
The purpose of this study is to assess the relative bioavailability by measuring the extent and rate of absorption of different tablet formulations of AZD1656 in T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Males or females of non-childbearing potential (post-menopausal, and/or have undergone hysterectomy and/or bilateral oophorectomy or salpingectomy/ tubal ligation) aged ≥18 years. Females will be defined as post-menopausal if last menstruation period was >1 year ago and serum follicle stimulating hormone (FSH) is within the post-menopausal range, or if age >50 years and with last menstruation period >2 years ago.
* A confirmed clinical diagnosis of T2DM for at least 1 year, treated with metformin as a single treatment or in combination with one other oral anti-diabetic (ie, DPPIV inhibitor or SU) for at least 2 months prior to screening. Doses of anti-diabetic treatment should have been stable for at least 1 month prior to screening.
* Treatment with at least 1000mg of Metformin for 2 months and being stable on the Metformin Therapy for 1 month
* Hb A1c >6.5% (international standard) at enrolment.
* Body mass index (BMI) between ≥19 and ≤42 kg/m2.

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the Investigator, within 2 weeks prior to the first administration of AZD1656
* Participation in another clinical study during the 30 days prior to screening or intake of another investigational drug within 30 days (or at least 5 x t1/2 of the drug) prior to the first administration of AZD1656.
* History of, or ongoing, ischemic heart disease or heart failure. Stroke, transitory ischemic attack, or symptomatic peripheral arterial disease within the last 6 months.
* Clinically significant abnormalities in ECG, clinical chemistry, hematology or urinalysis results.
* Positive test for Hepatitis B surface antigen (HBsAg) or antibodies to human immunodeficiency virus (HIV) or Hepatitis C virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of AUC of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 1
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of Cmax of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 1
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of tmax of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 1
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of AUC of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 2
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of Cmax of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 2
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of tmax of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 2
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of AUC of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 3
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of Cmax of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 3
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of tmax of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 3
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of AUC of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 4
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of Cmax of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 4
Measure: rate and extent of absorption of AZD1656 following single-dose administration of Tablets A, B, and C, administered before food intake and following administration of Tablet B after food intake, by assessment of tmax of AZD1656. | Blood samples will be collected from predose to 48 hrs at each treatment period 4

SECONDARY OUTCOMES:
To evaluate the safety of AZD1656 by assessing a panel of adverse events measures: physical examination, electrocardiogram, pulse and blood pressure, weight and laboratory, variables including plasma glucose. | start of treatment until follow up
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC | PK blood samples will be collected from predose to 48 hrs after each treatment period 1
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC(0-t). | PK blood samples will be collected from predose to 48 hrs after each treatment period 1
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of Cmax. | PK blood samples will be collected from predose to 48 hrs after each treatment period 1
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of tmax. | PK blood samples will be collected from predose to 48 hrs after each treatment period 1
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of t½. | PK blood samples will be collected from predose to 48 hrs after each treatment period 1
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC. | PK blood samples will be collected from predose to 48 hrs after each treatment period 2
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC(0-t). | PK blood samples will be collected from predose to 48 hrs after each treatment period 2
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of Cmax. | PK blood samples will be collected from predose to 48 hrs after each treatment period 2
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of tmax. | PK blood samples will be collected from predose to 48 hrs after each treatment period 2
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of t½. | PK blood samples will be collected from predose to 48 hrs after each treatment period 2
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC. | PK blood samples will be collected from predose to 48 hrs after each treatment period 3
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC(0-t). | PK blood samples will be collected from predose to 48 hrs after each treatment period 3
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of Cmax. | PK blood samples will be collected from predose to 48 hrs after each treatment period 3
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of tmax. | PK blood samples will be collected from predose to 48 hrs after each treatment period 3
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of t½. | PK blood samples will be collected from predose to 48 hrs after each treatment period 3
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC. | PK blood samples will be collected from predose to 48 hrs after each treatment period 4
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC(0-t). | PK blood samples will be collected from predose to 48 hrs after each treatment period 4
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of Cmax. | PK blood samples will be collected from predose to 48 hrs after each treatment period 4
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of tmax. | PK blood samples will be collected from predose to 48 hrs after each treatment period 4
Evaluate: pharmacokinetics of the AZD1656 metabolite, following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of t½. | PK blood samples will be collected from predose to 48 hrs after each treatment period 4
pharmacodynamics of AZD1656 following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC(0-4) and AUC(0-24) for glucose | PK blood samples will be collected from predose to 48 hrs after treatment period and P-glucose on Day 1 of each treatment period
pharmacodynamics of AZD1656 following single-dose administration of Tablets A, B, and C, given before food intake and following administration of Tablet B after food intake, by assessment of AUC(0-4) for insulin | PK blood samples will be collected from predose to 48 hrs after treatment period and P-glucose on Day 1 of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Eva Johnsson, MD, PhD, Study Director — AstraZeneca Sweden; Mark Matson, MD, Principal Investigator — Prism Research; Mirjana Kujacic Kujacic, MD, PhD, Study Chair — AstraZeneca R&D Mölndal
Locations (1):
- Research Site, Saint Paul, Minnesota, United States